CLINICAL TRIAL: NCT05047133
Title: Does Early Administration of Tranexamic Acid Decrease Perioperative Blood Loss in Addition to Intraoperative Tranexamic Acid for Hip Fracture Patients?
Brief Title: Effect of Early Administration of TXA in Adult Hip Fractures
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ascension Health (Industry)
Responsible Party: Principal Investigator, Jacob Hinkley, Resident Physician, Ascension Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1722787-1
Record Dates: First submitted 2021-09-03; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Postoperative Blood Loss
MeSH Terms: conditions — Postoperative Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Early Adminstration of TXA + Intraoperative TXA (Experimental): This group receives 1 G of TXA as soon as possible after a diagnosis of an acute hip fracture if the patient meets inclusion and exclusion criteria. The group will also receive 2 grams of TXA total intraoperatively.
  Interventions: Drug: Tranexamic acid
- Intraoperative only TXA (Other): This group will only receive the intraoperative TXA.
  Interventions: Drug: Tranexamic acid

INTERVENTIONS:
Drug: Tranexamic acid — TXA to be given at time of diagnosis in the emergency department (ED) in treatment group and at time of operation for both groups
  Other Names: Lysteda

SUMMARY:
This is a prospective clinical study designed to assess blood loss in intracapsular and extracapsular hip fractures undergoing operative fixation at a Level II trauma center. It is well established in the orthopedic literature that tranexamic acid (TXA) decreases blood loss and need for postoperative blood transfusion in hip fracture patients as well as total joint arthroplasty patients. A typical dosing pattern, and the dosing pattern employed at our institution, is 1 gram IV infused prior to incision followed by 1 gram IV infused at the time of wound closure.

ELIGIBILITY:
Inclusion Criteria:

* 1. All adult (18 years old or older) hip fracture patients presenting with an acute hip fracture and undergoing operative fixation

Exclusion Criteria:

1. Polytrauma patients
2. Previous operation on the ipsilateral hip
3. Patients with coagulopathies (Factor V Leiden, Sickle Cell Anemia, Etc.)
4. Patients with < 6-month history of thromboembolic event (DVT/PE), Stroke, Cardiac Stents, or Myocardial Infarction (MI)
5. History of seizure disorder
6. Patients on birth control
7. Pregnant Women
8. Prisoners
9. Active thromboembolic disease (DVT/PE, MI, Stroke)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Blood Transfusion | Up to two weeks
  Patient receives a blood transfusion during their postoperative stay in the hospital
Overall Blood Loss | Up to two weeks
  Calculate the difference in postoperative blood loss between groups

SECONDARY OUTCOMES:
Length of hospital stay | Up to two weeks
  Overall length of hospital stay
Postoperative Pain | Up to two weeks
  Difference in overall pain scores between groups
Wound complications | Up to two weeks
  Acute wound complications documented after surgical intervention
Acute DVT/PE | Up to two weeks
  Documented deep venous thrombosis or pulmonary embolism

CONTACTS AND LOCATIONS:
Locations (1):
- Ascension Genesys Hospital, Grand Blanc, Michigan, United States

IPD SHARING:
Plan to Share IPD: No